CLINICAL TRIAL: NCT03330756
Title: The Effects of the Laparoscopic Roux-en-Y Gastric Bypass and the Laparoscopic Mini Gastric Bypass on the Remission of Type II Diabetes Mellitus and the Pathophysiological Mechanisms That Drive the Conversion of Malign to Benign Obesity
Brief Title: The Effects of the Laparoscopic Roux-en-Y Gastric Bypass and Laparoscopic Mini Gastric Bypass on the Remission of Type II Diabetes Mellitus
Acronym: DIABAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Slotervaart Hospital (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1729
Record Dates: First submitted 2017-10-13; First posted 2017-11-06 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Obesity, Morbid; Type 2 Diabetes Mellitus
Keywords: Roux-en-Y gastric bypass; Mini gastric bypass; Type 2 diabetes mellitus; Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Single-center, open randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Roux-en-Y gastric bypass (Active Comparator): Laparoscopic Roux-en-Y gastric bypass
  Interventions: Procedure: laparoscopic Roux-en-Y gastric bypass
- Laparoscopic Mini Gastric Bypass (Experimental): laparoscopic Mini gastric bypass
  Interventions: Procedure: laparoscopic Mini gastric bypass

INTERVENTIONS:
Procedure: laparoscopic Roux-en-Y gastric bypass — laparoscopic Roux-en-Y gastric bypass with a 50 cm biliary limb and a 150 cm alimentary limb
  Other Names: gastric bypass
  Arms: Laparoscopic Roux-en-Y gastric bypass
Procedure: laparoscopic Mini gastric bypass — laparoscopic Mini gastric bypass with a gastrojejunostomy at 200 centimeters measured from the ligament of Treitz
  Other Names: One anastomosis gastric bypass, omega loop gastric bypass
  Arms: Laparoscopic Mini Gastric Bypass

SUMMARY:
It is estimated that there will be 439-552 million people with type 2 diabetes mellitus (T2DM) globally in 2030. Type 2 Diabetes Mellitus is present in one quarter of patients at the bariatric outpatient clinic. It is undecided which metabolic surgery grants best results in the remission of T2DM and which procedure does that at the lowest rate of surgical complications, long term difficulties and side effects. Non alcoholic fatty liver disease (NAFLD) is present in 80% of all morbidly obese subjects and is a major risk factor for development of insulin resistance and non alcoholic steatohepatis (NASH). It is increasingly recognized that the immune system, possibly driven by innate lymphoid cells (ILC's), and the intestinal microbiome are major players in this obesity related disease and the switch from benign to malign (insulin resistance and T2DM) obesity. However, the exact mechanisms of action behind the surgery-driven switch back from malign to benign obesity are unknown.Primary objective is to evaluate and compare the glycaemic control in T2DM within the first year of LRYGB and LMBG. Secondary aim is to gain insight in the pathophysiological mechanisms that drive the conversion of malign to benign obesity.

DETAILED DESCRIPTION:
Metabolic surgery has proven to be a viable long-term solution in the treatment of morbid obesity and its comorbidities. It induces rapid remission of type 2 diabetes mellitus (T2DM). Type 2 Diabetes Mellitus is present in one quarter of patients at the bariatric outpatient clinic. Non alcoholic fatty liver disease (NAFLD) is present in 80% of all morbidly obese subjects and is a major risk factor for development of insulin resistance and non alcoholic steatohepatis (NASH), with the latter becoming the major indication for liver transplantation in the USA. It is increasingly recognized that the immune system, possibly driven by innate lymphoid cells (ILC's), and the intestinal microbiome are major players in this obesity related disease and the switch from benign to malign (insulin resistance and T2DM) obesity. However, the exact mechanisms of action behind the surgery-driven switch back from malign to benign obesity are unknown. Also, it is undecided which metabolic surgery grants best results in the remission of T2DM and which procedure does that at the lowest rate of surgical complications, long term difficulties and side effects. The Laparoscopic Roux-en-Y Gastric Bypass (LRYGB), an efficient but complex procedure, is the golden standard in the Netherlands. The Laparoscopic Mini Gastric Bypass (LMGB) is technically less challenging and has been introduced to overcome some of the limitations of LRYGB. It has been hypothesized that the LMGB has a more rapid and durable glycaemic control, possibly due to the altered constitution and the augmented length of the biliary limb. There is reason to believe that the improved glycaemic control might become apparent within the first year of surgery and that it might remain thereafter. However, it is unknown what order of magnitude is to be expected and whether subgroups of T2DM patients will benefit the LMGB more. Also, it is unknown whether and to what extent intestinal microbiota and immunological tone can predict the metabolic response (improvement in insulin sensitivity) and NAFLD/NASH reduction and whether differences are expected between these two surgeries. Increased understanding of the pathophysiological mechanisms as well as their relationship to metabolic disturbances are thought to be of crucial importance to discover new diagnostic and therapeutical targets in obesity associated insulin resistance/T2DM and NAFLD/NASH. Primary objective is to evaluate and compare the glycaemic control in T2DM within the first year of LRYGB and LMBG. Secondary aim is to gain insight in the pathophysiological mechanisms that drive the conversion of malign to benign obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥35 and ≤50 kg/m2
* Diagnosis and treatment of T2DM at intake at bariatric ward with use of anti-diabetic medication.
* American Society of Anaesthesiologist Classification (ASA) ≤3
* All patients are required to lose 6 kilograms of weight prior to surgery

Exclusion Criteria:

* Known genetic basis for insulin resistance or glucose intolerance
* Type 1 DM
* Prior Bariatric surgery
* Patients requiring a concomitant intervention (such as cholecystectomy, ventral hernia repair)
* Auto-immune gastritis
* Known presence of gastro-esophageal reflux disease
* Known presence of large hiatal hernia requiring concomitant surgical repair
* Coagulation disorders (PT time > 14 seconds, aPTT ((dependent on laboratory methods) or known presence of bleeding disorders (anamnestic))
* Known presence of hemoglobinopathy
* Uncontrolled hypertension (RR > 150/95 mmHg)
* Renal insufficiency (creatinine > 150 umol/L)
* Pregnancy
* Breastfeeding
* Alcohol or drug dependency
* Primary lipid disorder
* Participation in any other (therapeutic) study that may influence primary or secondary outcomes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
glycaemic control | 12 months FU
  as measured by the difference in HBa1C

SECONDARY OUTCOMES:
glycaemic control | 6 and 24 months FU
  as measured by the difference in HBa1C
glycaemic control | 6, 12 and 24 months FU
  as measured by the difference in HBa1C and anti-diabetic medication
Insulin sensitivity | baseline, 12, 24 months FU
  Mixed meal tolerance test for level of insulin sensitivity
NAFLD/NASH | day of surgery, reoperation
  NAFLD/NASH parameters in liver biopsy measured with the Steatosis, Activity and Fibrosis (SAF) score according to Bedossa et al (2012).For each patient a SAF score summarizing the main histological lesions will be defined. The steatosis score (S) will assess the quantities of larger or median-sized lipid droplets but not foamy microvesicules from 0 to 3 (S0 <5%; S1 5-33%; S2 34-66% and S3>67%). Activity grade (A) from 0-4 is the unweighted addition of hepatocyte ballooning (0-2) and lobular inflammation (0-2). Stage of fibrosis will be assessed using the score described by NASH-CRN as follows; stage 0 (F0) no fibrosis; stage 1 (F1) 1a or 1b perisinusoidal zone 3 or 1c portal fibrosis; stage 2 (F2) persinusoidal and periportal fibrosis without bridging; stage 3 (F3) bridging fibrosis and stage 4 (F4) cirrhosis. A diagnostic algorithm which will be used during this study can be found in the original paper published by Bedossa et al.
Presence of bacterial DNA/bacterial metabolites - portal vein | day of surgery, reoperation
  in portal vein blood
Presence of bacterial DNA/bacterial metabolites - liver | day of surgery, reoperation
  in liver
Presence of bacterial DNA/bacterial metabolites - abdominal adipose tissue | day of surgery, reoperation
  in abdominal adipose tissue depots
Expression and differentiation of intestinal immunological cells - GALT | day of surgery, reoperation
  in GALT
Expression and differentiation of intestinal immunological cells - abdominal adipose tissue | day of surgery, reoperation
  in abdominal adipose tissue depots
Expression and differentiation of intestinal immunological cells - liver | day of surgery, reoperation
  in liver
Expression and differentiation of intestinal immunological cells - peripheral blood | day of surgery, reoperation
  in peripheral blood
Expression and differentiation of immunological cells | 12 and 24 months FU
  ILC's, macrophages
Expression and differentiation of inflammatory markers | 12 and 24 months FU
  IL6, IRX3 and 5
Small intestinal and fecal microbiota composition | 2, and 6 weeks, 6 months, as well as 12 and 24 months after surgery
  feces
Peripheral blood inflammatory markers | 2, and 6 weeks, 6 months, as well as 12 and 24 months after surgery
  ILC's, macrophages, T/B-cells and dendritic cells
Eating habits | baseline, 12, 24 months FU
  G-food craving questionnaire (FCQ-T) 21 item questionaire scale 0 (never) - 6 (always)
Eating habits | baseline, 12, 24 months FU
  10 questions, scale 0-10 for instance 0 not hungry -10 very hungry / satiety / craving salty food / craving sweet food / craving fat food
Excreted metabolites | baseline, 12, 24 months FU
  urine
Bio electric impedance | baseline, 12, 24 months FU
  body composition as assesed by bioelectical impedance analysis (BIA): the measurement of body fat in relation to lean body mass.
Quality of life | baseline, 12, 24 months FU
  Quality of life (IWQOL lite) 5 domain questionaire, 31 items: 1 never true - 5 always true
Cardiac / ventricular hypertrophy | baseline, 12, 24 months FU
  Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Maurits de Brauw, MD PhD, Principal Investigator — Head of department of Surgery
Locations (1):
- medical Center Slotervaart, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pyykko JE, Hinnen C, Aydin O, Nieuwdorp M, De Brauw LM, Bruin SC, van Olst N, Gerdes VEA, Sanderman R, Hagedoorn M. Attachment style and post-bariatric surgery health behaviours: the mediating role of self-esteem and health self-efficacy. BMC Psychol. 2023 Aug 25;11(1):248. doi: 10.1186/s40359-023-01273-5. PMID 37626349
- [Derived] van Rijswijk A, van Olst N, Meijnikman AS, Acherman YIZ, Bruin SC, van de Laar AW, van Olden CC, Aydin O, Borger H, Beuers UHW, Herrema H, Verheij J, Apers JA, Backhed F, Gerdes VEA, Nieuwdorp M, de Brauw LM. The effects of laparoscopic Roux-en-Y gastric bypass and one-anastomosis gastric bypass on glycemic control and remission of type 2 diabetes mellitus: study protocol for a multi-center randomized controlled trial (the DIABAR-trial). Trials. 2022 Oct 22;23(1):900. doi: 10.1186/s13063-022-06762-3. PMID 36273149